CLINICAL TRIAL: NCT00078052
Title: Genetic Markers of Coronary Heart Disease in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank B. Hu, Professor, Harvard School of Public Health (HSPH)
Other Study IDs: 1236; 5R01HL071981-04 (NIH)
Record Dates: First submitted 2004-02-17; First posted 2004-02-19 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus, Non-insulin Dependent; Diabetes Mellitus; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat

SUMMARY:
To investigate genetic markers of coronary heart disease in type 2 diabetes.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD), as the leading cause of death in the United States, is of significant public health concern. Despite the knowledge that atherosclerosis is the underlying cause of CHD, the recognition that both genetic and environmental factors contribute to the occurrence of disease, and the identification of a large number of genetic and environmental factors that have been found to be associated with disease risk, the etiology of atherosclerosis with the later development CHD continues to be not very well understood.

DESIGN NARRATIVE:

The nested case-control study will determine whether variability in 20 genes belonging to endothelial and inflammatory dysfunction pathways is related to the risk of coronary heart disease (CHD) among men and women diagnosed with type 2 diabetes in two large ongoing prospective studies, the Nurses' Health Study (NHS) and Health Professionals' Follow-up Study (HPFS). This will be accomplished by combining two complementary approaches that are made possible by the recent advances in knowledge of the human genome and high-throughput genotyping technologies. The investigators will directly target functional variants in the coding regions of the candidate genes and also investigate the association between CHD and ancestral haplotypes at each locus. The specific aims are: 1. To identify novel variants in 10 candidate genes of the inflammatory, and endothelial dysfunction pathways that have not been systematically screened for polymorphisms by targeted resequencing; 2. To assess the relationship between functional variants in 20 candidate genes in the inflammatory and endothelial dysfunction pathways and risk of CHD among subjects with diabetes of the NHS and HPFS cohorts; 3. To identify the subset of polymorphisms that best capture the overall genetic variability at each locus (haplotype tagging single nucleotide polymorphisms (SNPs) or htSNPs) and investigate the association between CHD risk and the haplotypes defined by these htSNPs; 4. To examine individual SNPs as well as haplotypes in relation to biochemical markers of inflammation and endothelial activation such as CRP, ICAM-1, VCAM-1, E-selectin, and TNF-a in diabetic individuals; and 5. To examine gene-environment interactions in relation to CHD risk in diabetic subjects. By 2006, an estimated 820 cases of CHD will have been confirmed among diabetic men and women in the blood cohorts. The large size, prospective design, high follow-up rates, detailed and reliable long-term lifestyle and outcome information, and the availability of blood specimens make these cohorts a valuable and unique resource for studying genetic determinants of accelerated atherosclerosis in diabetic patients.

ELIGIBILITY:
no history of CVD or cancer at baseline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nurses' Health Study and Health Professionals' Follow-up Study
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Actual)
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
cardiovascular disease | 1990-2006

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hu, Principal Investigator — Harvard School of Public Health (HSPH)

REFERENCES:
- [Background] Ma X, Bacci S, Mlynarski W, Gottardo L, Soccio T, Menzaghi C, Iori E, Lager RA, Shroff AR, Gervino EV, Nesto RW, Johnstone MT, Abumrad NA, Avogaro A, Trischitta V, Doria A. A common haplotype at the CD36 locus is associated with high free fatty acid levels and increased cardiovascular risk in Caucasians. Hum Mol Genet. 2004 Oct 1;13(19):2197-205. doi: 10.1093/hmg/ddh233. Epub 2004 Jul 28. PMID 15282206